CLINICAL TRIAL: NCT05602181
Title: Effects of the Accessible Literacy Learning (ALL) App on Early Literacy Skills by Children Who Use Augmentative and Alternative Communication
Brief Title: Effect of the ALL App on Literacy for Children Who Use AAC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Jessica Caron, Assistant Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00018772
Record Dates: First submitted 2022-10-10; First posted 2022-11-01 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Literacy
Keywords: AAC
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ALL Phonics Instruction (Experimental): Lessons for the treatment group will be 30-min. long using the ALL app with a known service provider. Lessons will include systematic instruction with four subskills per session (e.g., letter-sounds, sound blending, typing, and sight words). The words and subskills with rotate based on the data collected and the machine learning within the technology. The child will complete 100 lessons. The systematic instruction with subksills (e.g., sound blending, decoding) includes 10 trials per word and an instructional sequence that introduces the skill, two models, six trials of guided practice, and two trials of independent practice with corrective feedback.
  Interventions: Behavioral: ALL Phonics Instruction
- ALL Sight Word (Active Comparator): Lessons for the comparison group will be 30-min. long using the ALL app with a known service provider. Lessons will include systematic instruction with sight words. The child will also complete 100 lessons.No phonics instruction will be provided to this group through the ALL app.
  Interventions: Behavioral: ALL Sight Word Instruction

INTERVENTIONS:
Behavioral: ALL Phonics Instruction — The Accessible Literacy Learning (ALL) App is available in the app store and created by TobiiDynavox (an AAC device company). The ALL app is evidence informed and includes pre-made lessons in early phonics/phonological skills including: letter-sounds, sound blending, decoding, phoneme segmentation, sight words, and encoding. The materials made in the app are adapted and created for children with minimal or no speech.
  Arms: ALL Phonics Instruction
Behavioral: ALL Sight Word Instruction — The Accessible Literacy Learning (ALL) App is available in the app store and created by TobiiDynavox (an AAC device company). The ALL app is evidence informed and includes pre-made lessons in early phonics/phonological skills including: letter-sounds, sound blending, decoding, phoneme segmentation, sight words, and encoding. The materials made in the app are adapted and created for children with minimal or no speech. This group will only use the sight word lessons, as well as the library for sight word books. No phonics instruction will be provided through the app.
  Arms: ALL Sight Word

SUMMARY:
The goal of this clinical trial is to test a phonics-based literacy program for children with limited or no speech who use augmentative and alternative communication.

More specifically, this study aims to:

1. Understand if using a literacy app (Accessible Literacy Learning) created to support individuals with limited or no speech, with instruction provided by a service provider, will increase their literacy skills
2. Understand how many trials/how much time it takes to acquire each of the 6 early literacy skill assessed
3. Understand if service providers think the Accessible Literacy Learning app is appropriate for this population that needs many literacy adaptions due to challenges with speech.
4. Understand if any characteristics lead to more learning of the skills, for example, diagnosis or age

Participants will be asked to complete 100 lessons using the app. The lessons will be phonics-based for the intervention group. The comparison group with use the same app and complete 100 lessons, but will only complete lessons in sight word (no phonics).

ELIGIBILITY:
Inclusion Criteria:

Students with CCN can participate if they meet the following criteria:

* 3 to 10 years old
* present with speech and communication skills that did not meet all of their daily communication needs (e.g., have an AAC system; less than 50% intelligible at the single word level to unfamiliar partners if using speech)
* follow one-step directions
* symbolic communicators with use of at least 50 words/signs/picture icons expressively,
* limited literacy skills (i.e., identify less than 26 letter-sound correspondences, 10 words during sound blending, 25 sight words on the screening assessment, and can spell less that 20 words)
* not receiving consistent phonologically-based direct literacy instruction or receiving instruction in less than 2 of the tested skills
* unimpaired or corrected vision and hearing
* access to an iPad

School support personnel (e.g., teachers, speech-pathologists, paraprofessionals) can participate if they meet the following criteria, per self-report:

* Speaks English
* Reads English
* 18 years of age or older
* Spending time directly working with an individual with CCN who needs to learn to read
* Willingness to implement the ALL curriculum and incorporate it into the daily educational plans

Exclusion Criteria:

Students cannot participate if they:

* are under 3 years of age
* do not present with severe speech disorders whereby they could use or benefit from AAC
* can't follow one-step directions
* are not symbolic communicators
* are able to read at the connected text level
* do not speak/understand English
* impaired and uncorrected vision and hearing
* do not have access to an iPad to use the ALL app

Support personnel cannot participate if they:

* do not speak English
* do not understand English
* have impaired vision and hearing that is not corrected and impacts reading and hearing the child they work with
* are not in daily direct contact with someone with CCN
* unwilling to attend trainings related to the ALL app
* unwilling to incorporate the ALL app into daily educational plans

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Scores on the Early Literacy Assessment | Through study completion, an average of 8 months
  We will examine the impact of literacy lessons delivered with the ALL technology on the change in scores on the Early Literacy Assessment (ELA) -specifically change in scores in the areas of letter-sounds, sound blending, phoneme segmentation, decoding, irregular sight words, and encoding.

SECONDARY OUTCOMES:
Data from the Feasibility Adoption Acceptability Questionnaire (FAAQ) | Through study completion, an average of 8 months
  To measure the perceptions of implementation variables the Feasibility Adoption Acceptability Questionnaire (FAAQ) will be completed at six timepoints throughout the study. Likert-scale questions (Scale of 1-5) across 10 questions, as well as 2 open responses.
Treatment and Acceptability Rating Form - Revised | Through study completion, an average of 8 months
  Pre-post interviews using the Treatment and Acceptability Rating Form-Revised (TARF-R) [20] will examine which components of the ALL technology are perceived as helpful or hindering to progress as well as factors that may support high implementation fidelity.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Caron, Ph.D., Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennsylvania State University, State College, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographic information, as well as raw scores on literacy assessment measures.
Time Frame: After analysis of results (approximately November 2025)